# **Evaluation of Smell and Taste in Fibromyalgia- NCT03823937**

## 06/01/2019

#### **Study Protocol:**

#### **Participants**

18-70 years old consecutive FM patients diagnosed according to ACR criteria 2016 revision and age, sex-matched healthy controls were included in the study. Neurologic disorders, rheumatologic and endocrine diseases, diabetes mellitus, traumatic brain injury, psychiatric disorders, chronic rhinitis/sinusitis/rhinosinusitis, history of head trauma or operation, malignancies, and pregnancy were defined as exclusion criteria. Besides, patients taking any antidepressants, pregabalin or gabapentin were excluded from the study.

According to ACR criteria 2016 revision criteria widespread pain index (WPI), symptom severity scale (SSS) score and fibromyalgia severity scale (FSS) score which is the sum of WPI and SSS was calculated. Fibromyalgia impact questionnaire (FIQ) which measures patient status was applied to FM patients. EuroQol Questionnaire 5-Dimensions (EQ-5D) was applied to all participants to assess QoL. Hamilton anxiety and depression scale were administered by the psychiatrist who is unaware of the diagnosis. Toronto Alexithymia Scale (TAS-20) was used for measurement of alexithymia which refers to trouble in identifying and describing emotions.

Sniffin' Sticks test which consists of odor threshold (T), discrimination (D) and identification (I) subtests was used. Taste strips taste (Brughart Medical Technology, Wedel, Germany) which consists of 16 filter paper taste strips was used.

### **Statistical Analysis:**

The IBM SPSS Statistics 22 (SPSS IBM, Turkey) program was used for statistical analysis. The normality of the parameters was assessed with the Shapiro-Wilk test. Mean, median, standard deviation, and frequency was used as descriptive statistical methods. The Student's t-test was used to make comparisons between the parameters in each group that showed normal distribution, and the Mann-Whitney U test was used to make comparisons between the parameters in each group that lacked normal distribution. The chi-square test, Fisher's exact test, and Yates continuity correction were used to compare the qualitative data. For the analysis of the correlation between the parameters, Spearman test was performed. Significance was assessed at p<0.05 level, 95% confidence interval.